CLINICAL TRIAL: NCT05220592
Title: Learning How to Recover From Stress: Results From an Internet-based Randomized Controlled Pilot Trial
Brief Title: Learning How to Recover From Stress - Pilot RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: iStress4
Record Dates: First submitted 2022-01-20; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Adjustment Disorders
Keywords: Recovery; Stress; Internet-based; Prevention; Intervention; Work
MeSH Terms: conditions — Adjustment Disorders

STUDY DESIGN:
Intervention Model Description: This study was a two-armed controlled trial in which an internet-based recovery training program (iRTP) was compared with a wait-list control group (WLC). The study followed Consolidated Standards of Reporting Trials (CONSORT) guidelines (Schulz et al., 2010) and was conducted between February 2018 and May 2019. Since this was a pilot trial, no power calculation and estimates of sample size were conducted.
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based recovery training program (n=35) (Experimental): The iRTP was based on recovery experiences (psychological detachment, relaxation, mastery, and control), converted into a recovery training intervention inspired by Hahn et al. (2011). The iRTP comprised five modules distributed over five weeks, with modules lasting 60-120 minutes per week.
  Interventions: Behavioral: Internet-based recovery training program
- Wait-list control group (n=34) (No Intervention): Wait-list control group received equal and parallell assessment and eligibility procedure as the experimental conditions. Wait-list control group gained access to iCBT/W-iCBT program after the six months follow-up.

INTERVENTIONS:
Behavioral: Internet-based recovery training program — The iRTP was based on recovery experiences (psychological detachment, relaxation, mastery, and control), converted into a recovery training intervention, and inspired by Hahn et al. (2011). The iRTP comprised five modules distributed over five weeks, with modules lasting 60-120 minutes per week. Each module contained psycho education, worksheets, images, cases, audio and video files, and homework assignments.
  Arms: Internet-based recovery training program (n=35)

SUMMARY:
This randomized, controlled pilot trial evaluated the efficacy of a brief internet-based recovery training intervention targeting distressed employees. This pilot trial is one of the first to examine a brief recovery training program's efficacy, suggesting that employees across a wide range of professions could learn how to recover from elevated stress symptoms. This type of accessible and brief recovery intervention might shape the future of stress prevention, but more research is needed with larger samples before further conclusions can be drawn.

DETAILED DESCRIPTION:
In recent years, work-related stress and burnout have received more attention, with a higher prevalence observed within the working population. Today, every fourth employee has experienced stress during most of their working days. Employees exposed to prolonged stress in their work situations experience more strain and suffer from poor well-being; higher risk of severe health implications, such as coronary artery disease; and problems in work participation, such as sickness absences, including long-term sick leave.

Empirical research suggests that recovery from work is important in reducing the negative effects on employees from stress and strain, as well as preserving their well-being and work performance. Recovery refers to the restoration processes during which a person's stress level returns to its pre-stress level. Recovery as a process refers to the activities and experiences that elicit change in stress and strain indicators. Recovery as an outcome captures a person's psychological or physiological state reached after a recovery period (e.g., at the end of a workday). Confirmatory factor analysis has proposed four distinct experiences in recovering from work processes: psychological detachment; relaxation; mastery; and control. Extant studies confirm that these experiences are related positively to well-being indicators such as the Recovery Experience Questionnaire.

Although extensive research has been devoted to stress intervention programs, and evidence suggest that these are effective in reducing stress within the working population, few studies have evaluated interventions aimed at stress prevention, e.g., by removing stressors and/or enhancing well-being factors, such as recovery. Most stress interventions have focused on reducing participants' cognitive, emotional, and behavioral symptoms when coping with stress. However, some promising results on stress prevention have been observed from recovery training programs.

Despite the evidence on the efficacy of stress management interventions and some promising results from recovery training interventions , only a small percentage of distressed employees actually receive stress interventions. This calls for further development and evaluation of interventions that are accessible and has the potential in preventing chronic stress in the working population.

The internet has the potential to disseminate interventions broadly, and a growing body of literature has demonstrated internet-based stress interventions' efficacy, with small to moderate effects on outcomes from stress, burnout, insomnia, depression, and anxiety.

The present, controlled pilot study aim to examine the efficacy of a brief, five-week, internet-based recovery training program for employees experiencing elevated symptoms of stress and/or a stress-related disorder burnout in a randomized, controlled pilot trial. We hypothesize that the internet-based recovery program would produce greater improvements in recovery experiences (primary outcome) compared with a wait-list control group. We also hypothesize that the intervention group will differ with regard to important health-related (perceived stress, burnout, exhaustion, depression, alcohol consumption, and quality of life) and work-related (work experience, work ability, sickness absences) outcomes. Finally, we investigate whether the initially achieved changes in the intervention group would remain stable at six- and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

All participants were volunteers. To be eligible for the study, each participant had to fulfill the following criteria:

* at least 18 years old; (ii) fluent in Swedish
* have access to a computer or handheld device with internet access
* currently be employed
* >14 points on the Perceived Stress Scale
* <5 points on the Shirom Melamed Burnout Questionnaire (SMBQ)
* <20 points on the Montgomery Åsberg Depression Rating Scale-Self-Rated (MADRS-S)
* <21 points on the Insomnia Severity Index (ISI)
* <14 points on the Alcohol Use Disorders Identification Test (AUDIT).

Exclusion Criteria:

Participants were excluded from the study if they:

* currently were in treatment for stress or burnout;
* currently were suffering from bipolar disorder, psychosis, post-traumatic stress disorder (PTSD), eating disorders, substance abuse, severe forms of depression, anxiety disorder or personality disorders as assessed in a telephone interview (MINI)
* suicidal ideation based on Item 9 on the MADRS-S.
* If on medication (e.g., antidepressants or sleep medication) this should be held constant medication constant during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Recovery Experiences Questionnaire | Pre; 5 weeks
  The 16-item Recovery Experience Questionnaire (REQ) includes four factors, representing four different recovery experiences; (i) psychological detachment (ii) relaxation, (iii) mastery and (iv) control. The questionnaire is answered on a 5-point Likert scale, and has been validated in a Swedish population showing excellent internal consistency, α=0.92 [83].

SECONDARY OUTCOMES:
Shirom-Melamed Burnout Questionnaire | Pre; 5 weeks
  The Shirom-Melamed Burnout Questionnaire (SMBQ), is a 22-item scale (graded 1-7) used to assess different aspects of chronic stress and burnout (Physical Fatigue, Cognitive weariness, Tension, and Listlessness). This scale correlates signiﬁcantly with other well established questionnaires measuring burnout, e.g., Maslach Burnout Inventory. The SMBQ has an internal consistency reliability (Cronbach's alpha) of .92..
Perceived Stress Scale | Pre; 5 weeks
  Perceived stress was measured with the 10-item version of the Perceived Stress Scale (PSS-14), translated into Swedish. The PSS-10 is designed to measure the degree to which situations in one's life are appraised as stressful. The Swedish version of PSS has an internal consistency reliability (Cronbach's alpha) of .82 and split-half reliability estimate of .84.
Karolinska Exhaustion Disorder Scale | Pre; 5 weeks
  Karolinska Exhaustion Disorder Scale (KEDS-9) is a 9-item questionnaire measuring symptoms of chronic stress, fatigue and exhaustion. The instrument is answered on a 7-point scale, with a scale range of 0-54. A cut-off score of 19 was shown to discriminate between healthy subjects and patients with chronic stress and exhaustion. KEDS-9 has satisfactory reliability, Cronbach's alpha of .94.
Montgomery Åsberg Depression Rating Scale | Pre; 5 weeks
  We used the Montgomery Åsberg Depression Rating Scale self-assessment, MADRS-S to measure symptoms of depression. MADRS-S consists of nine items measuring different symptoms of depression and each symptom is rated on a six-point scale. The instrument has good reliability and has been validated as an internet-based measure. In a comparative study the MADRS-S correlated highly (r = .87) with the Beck Depression Inventory, indicating acceptable convergent validity.
Generalised Anxiety Disorder Scale | Pre; 5 weeks
  Generalized Anxiety Disorder 7-item Scale (GAD-7) is an instrument assessing excessive worry and generalized anxiety disorder. GAD-7 had good internal consistency reliability (α = .83), test-retest reliability (r = .83), as well as criterion, construct, factorial, and procedural validity. A cut-off score of 10 has been suggested to discriminates between healthy subjects and patients with generalized anxiety disorder.
Insomnia Severity Index | Pre; 5 weeks
  The Insomnia Severity Index (ISI) is a 7-item self-report questionnaire that measures individuals perceptions of their insomnia and the severity of problems with delayed sleep onset, sleep maintenance, and early morning awakenings. ISI exhibits adequate internal consistency measures (α =.74), and is a sensitive measure to detect changes in perceived sleep difficulties. It has previously been validated as an internet-based measure.
Alcohol Use Disorders Identification Test | Pre; 5 weeks
  The Alcohol Use Disorders Identification Test (AUDIT) was used to assess potential alcohol dependence or abuse. In a study of the psychometric properties of the Swedish version of AUDIT, both internal and test-retest reliabilities were satisfactory. A cut-off of <14 points on the AUDIT indicating risk of overconsumption of alcohol.
Work Experience Measurement Scale | Pre; 5 weeks
  The Work Experience Measurement Scale (WEMS) is an instrument measuring the experience of work from a health resource perspective. WEMS consists of 32 items measuring job satisfaction in five different domains (supportive work conditions, internal work experience, autonomy, time experience, management, process of change) on a six-point scale. Cronbach's alpha on the WEMS has been reported to be in the interval of .85-.96.
Work Ability Index | Pre; 5 weeks
  Work Ability Index (WAI) is an instrument for assessing health status and work ability among employees. The WAI comprises of different scales, with scores ranging from 7 to 49 points. Studies have suggested that 7-27 points = poor; 28-36 points = moderate; 37-43 points = good; and 44-49 points indicates excellent work ability. Analyses of reliability indicates satisfactory internal consistency, α-levels ranging from .79 to .80.
International Physical Activity Questionnaire | Pre; 5 weeks
  The International Physical Activity Questionnaire (IPAQ) is a 10-item self-assessment questionnaire (short version) that aims to measure physical activity and inactivity. Participants are asked to rate all their physical activity (according to intensity level, e.g., walking, moderately strenuous activities, and very strenuous activities) and inactivity (i.e., sedentary time) in minutes over the previous seven days. The IPAQ has demonstrated acceptable reliability, test-retest reliability, and criterion validity (accelerometer) in various contexts and languages.
Brunnsviken Brief Quality of Life Inventory | Pre; 5 weeks
  The Brunnsviken Brief Quality of Life Inventory (BBQ) measures quality of life within six domains: self-respect; values; leisure time; learning; creativity; and friends. The instrument uses a five-point scale, with a scale range of 0-96. Each domain is assessed according to its importance and contentment. BBQ has satisfactory internal consistency reliability (α=.68) and test-retest reliability (r=.89).
Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry | Pre; 6 months
  TiC-P has been used in several studies for economic evaluations of healthcare consumption and productivity loss in mental health. Sickness absence were conceptualized as the self-rated number of days during the past three months absent from work while being physically or mentally ill.

OTHER OUTCOMES:
Recovery Experiences Questionnaire | 6-month, 12-month
  Primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Once published data will be made available on request via repository.
Time Frame: When published.
Access Criteria: On request or public.

REFERENCES:
- [Derived] Asplund RP, Carvallo F, Christensson H, Videsater E, Haggman A, Ljotsson B, Carlbring P, Andersson G. Learning how to recover from stress: Results from an internet-based randomized controlled pilot trial. Internet Interv. 2023 Oct 17;34:100681. doi: 10.1016/j.invent.2023.100681. eCollection 2023 Dec. PMID 38023967